CLINICAL TRIAL: NCT05732532
Title: Treatment of Headache With Occipital Nerve Blocks: Comparison Trial of Anesthetic With or Without Dexamethasone
Brief Title: Steroids in Occipital Nerve Block for Treatment of Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie (Beth) E. Robertson, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-007855
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Headache; Occipital Nerve Block
MeSH Terms: conditions — Headache | interventions — Bupivacaine; Lidocaine; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anesthetic without steroid group (Active Comparator): Subjects scheduled for bilateral greater/lesser occipital nerve blocks as part of clinical care will receive standard of care medication, including lidocaine and bupivacaine and normal saline.
  Interventions: Drug: Bupivacaine; Drug: Lidocaine; Drug: Normal saline; Procedure: Greater/lesser occipital nerve blocks
- Anesthetic with dexamethasone group (Experimental): Subjects scheduled for bilateral greater/lesser occipital nerve blocks as part of clinical care will receive standard of care medication, including lidocaine and bupivacaine and dexamethasone.
  Interventions: Drug: Bupivacaine; Drug: Lidocaine; Drug: Dexamethasone; Procedure: Greater/lesser occipital nerve blocks

INTERVENTIONS:
Drug: Bupivacaine — 2 mL of bupivacaine 0.5% (5 mg/mL) injected at the origin of each bilateral greater and lesser occipital nerves
Drug: Lidocaine — 0.5 mL of lidocaine 1% (10 mg/mL) injected at the origin of each bilateral greater and lesser occipital nerves
Drug: Dexamethasone — 0.5 mL of dexamethasone (10 mg/mL) injected at the origin of each bilateral greater and lesser occipital nerves
  Arms: Anesthetic with dexamethasone group
Drug: Normal saline — 0.5 mL of normal saline 0.9% injected at the origin of each bilateral greater and lesser occipital nerves
  Arms: Anesthetic without steroid group
Procedure: Greater/lesser occipital nerve blocks — Subjects will receive a total of 12 mL injectate divided equally between the 4 injection sites of the bilateral greater and lesser occipital nerves using the landmark-based technique.

SUMMARY:
Currently there is limited evidence of benefit for the addition of steroids to occipital nerve blocks for treatment of headache, and not all steroids have been explored. The purpose of this research is to learn more about whether the addition of a specific kind of steroid (dexamethasone) provides any additional benefit to nerve blocks.

DETAILED DESCRIPTION:
Patients who are referred by their neurology provider for occipital nerve block as treatment of headache according to current accepted standard of care will be considered for this study. Baseline data will be obtained from the patients prior to proceeding with their nerve block and their headache diagnosis will be recorded based on electronic medical record review. Patients will be randomized to one of two treatment arms, anesthetic with dexamethasone or anesthetic without dexamethasone. The injectate will be the same color and amount of solution for each trial arm. Thus, the neurology provider performing the injection remains blinded and the patient remains blinded.

Injection sites will be inspected to ensure no active bleeding, infection, cranial bone or cervical spine defects/prior surgeries that prohibit safe use of landmark-based technique. A neurologist who is experienced at performing nerve blocks will administer the injections to the bilateral greater and lesser occipital nerves using the landmark-based technique. The occipital protuberance and mastoid process are palpated, with the location of the greater occipital nerve at approximately 1/3 the distance laterally and the lesser occipital nerve at approximately 2/3 the distance laterally along the nuchal ridge for a total of 4 injection sites.

Patients will be observed for approximately 10 minutes after the procedure to monitor for any immediate adverse effects and to ensure that anesthesia in the distribution of the injected nerves was achieved. Then, they will be instructed to keep a headache diary after treatment and will be provided a written example diary. A study staff who remains blinded to the patient's trial arm (but not necessarily the neurology provider who performed the injection) will contact the patients via telephone at 1, 2 and 4 weeks to assess response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treated for headache including but not limited to occipital neuralgia, episodic migraine, chronic migraine and/or cervicogenic headache.
* Stable on preventative medication dosing for at least 1 month prior to occipital nerve block and no change in preventative medication regimen during the course of the study.
* Able to understand the requirements of the study and return for treatment.
* Able to independently provide informed consent.

Exclusion Criteria:

* Diagnosis of cluster headache according to the International Classification of Headache Disorders 3rd edition.
* Occipital or other cranial nerve block administered within 3 months prior to initiation of study.
* History of adverse reaction or contraindication to any of the study ingredients (bupivacaine, lidocaine, dexamethasone).
* Pregnancy.
* Infection or bleeding at site of injection.
* Cranial bone or cervical spine defects/prior surgeries near injection site that prohibit use of landmark-based technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Headache days 1 week following treatment | 1 week
  Number of self-reported days subjects experience headaches in the past week following treatment
Headache days 2 weeks following treatment | 2 weeks
  Number of self-reported days subjects experience headaches in the past weeks following treatment
Headache days 4 weeks following treatment | 4 weeks
  Number of self-reported days subjects experience headaches in the past weeks following treatment

SECONDARY OUTCOMES:
Headache Severity | 1 week, 2 weeks, 4 weeks
  Self-reported average severity of subjects' headaches using a scale of 0-10, with 0=no pain and 10=worst pain possible following treatment
Moderate or severe headache days | 1 week, 2 weeks, 4 weeks
  Number of self-reported days subjects report headaches as being moderate or severe following treatment
Acute medication use | 1 week, 2 weeks, 4 weeks
  Number of self-reported days subject had to take acute pain medication for their headaches following treatment
Location of headache | 1 week, 2 weeks, 4 weeks
  Self-reported location of headache (front, back, other) following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Robertson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No